CLINICAL TRIAL: NCT04105829
Title: Effects of the Different Orthodontic Fixed Retainers on Enamel Colour Change
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Aysegul Gulec, Principal investigator, University of Gaziantep
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 210
Record Dates: First submitted 2019-09-19; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Tooth Color
Keywords: tooth color change
MeSH Terms: interventions — RIBBOND

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tooth color measurement (Experimental): Tooth color changes between times (before retainer bonding, after retainer bonding, in 1 month, 3 months, 6 months and a year)
  Interventions: Other: Bond-a braid; Other: EverStick-Ortho; Other: Ribbond

INTERVENTIONS:
Other: Bond-a braid — Stainless steel lingual retainer application
Other: EverStick-Ortho — Fiber reinforced lingual retainer
Other: Ribbond — Fiber reinforced lingual retainer

SUMMARY:
The aim of this study is to compare the tooth colour changes caused by retainers made of stainless steel wires and fiber reinforced in long term

DETAILED DESCRIPTION:
30 patients who were planned to use lower fixed retainer after fixed orthodontic treatment, were included in the study and divided into 3 groups. (n=10) (Group 1: Bond a braid retainer, Group 2: Ribbond retainer, Group 3: EverStick Ortho retainer). Colour measurements will be made with spectrophotometer (Vita easyshade) after debonding (T1), after retainer application (T2), in 1 month, 3 month, 6 month and finally 1 year from 6 lower anterior teeth. The Commission Internationale de I'Echairage L*a*b* system will be used to determine the tooth colour. ∆E values measured at different times will be compared.

ELIGIBILITY:
Inclusion Criteria:

* patients with no anomalies of lower incisors and canine teeth

Exclusion Criteria:

* patients drinking more then 3 cups of coffee per day
* smoker patients

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2020-02-20 (Estimated)

PRIMARY OUTCOMES:
Tooth color change | before debonding, after debonding on 1st, 3rd, 6th months and 1st year
  Measurement of tooth color change with spectrophotometry

CONTACTS AND LOCATIONS:
Overall Officials: Merve Goymen, PhD, Study Chair — University of Gaziantep; Derya Sürmelioğlu, Study Chair — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No